CLINICAL TRIAL: NCT03817047
Title: A Cluster-randomized Controlled Trial Evaluating the Effect of Increased Physical Education and Physical Activity on Adolescents' Physical and Mental Health, Academic Performance and Learning Environment
Brief Title: The Effect of Increased Physical Activity on Adolescents' Health and Academic Performance: The School in Motion Study
Acronym: ScIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: University of Stavanger (Other); University of Agder (Other); Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Elin Kolle, Vice rector, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2207ScIM
Record Dates: First submitted 2019-01-14; First posted 2019-01-25 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Physical Activity; Academic Achievement; Mental Health
Keywords: Adolescents; Physical activity; Physical fitness; Academic performance; Cluster RCT; Mental health; Secondary school; Physical education; Physical active educational lessons; Accelerometer
MeSH Terms: conditions — Motor Activity; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized trial with three parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical active learning (PAL) (Experimental): Three components:
  1. Physical education (60 minutes)
  2. Physical active learning (30 minutes)
  3. Physical activity (30 minutes)
  Interventions: Behavioral: Physical education; Behavioral: Physical active learning; Behavioral: Physical activity
- Don't worry - be happy (Experimental): Two components:
  1. Physical education (60 minutes) - don't worry class
  2. Physical activity (60 minutes) - be happy class
  Interventions: Behavioral: Physical education; Behavioral: Be happy
- Control group (No Intervention): Current practice

INTERVENTIONS:
Behavioral: Physical education — Physical education (60 minutes): In addition to the ordinary PE-lessons. The pedagogical activities taught in this lesson should be in line with the curriculum of 9th grade and led by the PE-teacher. In the Don't worry - be happy intervention this class was also organized by the students. The students practiced their Be Happy-activities, or they introduced their class peers to their "Be Happy"-activity. A PE-teacher was present to support the students if necessary.
  Other Names: PE-intervention
  Arms: Don't worry - be happy; Physical active learning (PAL)
Behavioral: Physical active learning — The curriculum of the subjects (i.e. maths, English, Norwegian) were taught in a physically active manner. The lesson should last 30 minutes and be led by the teacher of the current subject.
  Arms: Physical active learning (PAL)
Behavioral: Physical activity — Without a connection to any specific subject "Physical activity" should be performed as 30 minutes a week. There are no specific aims to be taught in this lesson, but physical activities that stimulates mastery, joy and well-being should be in focus.
  Arms: Physical active learning (PAL)
Behavioral: Be happy — The Be Happy classes were self-organized activity groups of at least three students, developed according to activity preferences across regular classes. The Be Happy groups practiced traditional sports and physical activities, lifestyle sports, dancing, out-door recreation, drama etc. - inside or outside school.
  Arms: Don't worry - be happy

SUMMARY:
This study evaluates the effect of 120 minutes extra of physical education (PE) or physical activity (PA) on adolescents' physical health, mental health, academic performance and learning environment. This is a cluster-randomized controlled trial with three arms, where the participants in two of the groups will have different models of increased PE/PA during the school week, whereas the participants in the third arm is the control group including current practice.

DETAILED DESCRIPTION:
This is a school-based, three-arm cluster randomized controlled trial (RCT) recruiting adolescents from secondary schools in Norway. Adolescents (aged 14-15 years) were the unit of analysis, and schools (clusters) were randomly assigned to one of three conditions:

1. the physical active learning group (PAL-group), where the schools each week include one additional physical education (PE) lesson, 30 minutes of physical active learning, and 30 minutes of physical activity (intervention condition);
2. the don't worry - be happy group (DWBH-group), where the schools include one new activity class (60 minutes: Be Happy class) and one additional PE-class (60 minutes: Don't Worry class) per week (intervention condition);or
3. current practice (control condition). An identical set of outcome measures are taken from all participants at baseline, and approximately 12 months after the baseline measures, when the participants were at the end of year 9

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in 9th grade

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2045 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Mean physical activity level | Measured baseline and after 12 months
  The participants mean physical activity level measured by accelerometers

SECONDARY OUTCOMES:
Time spent in moderate-to-vigorous physical activity (MVPA) | Measured baseline and after 12 months
  Mean minutes spent in MVPA per day
Time spent sedentary | Measured baseline and after 12 months
  Mean minutes spent sedentary each day, measured both objectively using accelerometers
Sedentary behaviour | Measured baseline and after 12 months
  Self-reported in a questionnaire. There are questions related to minutes spent in front of a screen. The answers are categorized into seven alternatives ranging from "No time at all" to "More than 6 hours per day". There are also questions about which screen activity they perform. The answers are categorized into six alternatives ranging from "No time at all" to "More than 3 hours per day". There are also questions about time spent doing homework. The answers are categorized into nine alternatives ranging from "No time at all" to " More than 7 hours per day".
Upper limb strength | Measured baseline and after 12 months
  Handgrip strength using a hand dynamometer. The participants will use the dominant hand, with the arm completely extended and squeeze the dynamometer with maximum isometric effort, for about 2-3 seconds.
Explosive strength in the lower body | Measured baseline and after 12 months
  Standing broad jump. The participants will stand behind a line with feet slightly apart. They will be instructed to perform a two-foot take-off and landing, and to jump as far as possible, landing on both feet without falling backwards. The distance from the take-off line to the nearest point of contact on the landing (back of the heels) will be measured, and the better of two attempts will be used for analyses.
Abdominal muscle endurance | Measured baseline and after 12 months
  Abdominal muscular endurance will be measured by a sit-up test. The participant will start in a lying position with hands clasped behind the neck, knees bent at a 45° angle with the heels and feet flat on the floor and held down by the tester. The subject then rise to a position with the elbows pointed forward until they touched the knees. The total number of correctly performed and completed sit-ups within 30 seconds is counted.
Cardiorespiratory fitness | Measured baseline and after 12 months
  Intermittent running test. Participants run for 10 minutes, and the distance covered (in meters) is recorded.
Academic performance in reading | Measured baseline and after 9 months
  Specific standardized Norwegian National tests in reading.The test is designed and administrated by The Norwegian Directorate for Education and Training.
Academic performance in numeracy | Measured baseline and after 9 months
  Specific standardized Norwegian National tests in numeracy. The test is designed and administrated by The Norwegian Directorate for Education and Training.
Overall psychosocial problems and strengths | Measured baseline and after 12 months
  Assessed with the Strength and Difficulties Questionnaire (SDQ). This is a short screening instrument consisting of 25 items equally divided across five scales measuring emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior.
  Each statement is answered as "Not true", "Somewhat true" and "Certainly true". Some questions have reversed form, which is reversed in the scoring of the instrument. Replies were scored from 0 to 2, and the subscales are summed to a score ranging from 0-10 for each subscale. Added together, the first four scores generate a total difficulties score, ranging from 0 to 40. Higher scores indicate more problems.
Adolescents' subjective health and well-being | Measured baseline and after 12 months
  Adolescent's subjective health and well-being is assessed using the Kidscreen-27 questionnaire. The instrument consists of 27 items covering the following five quality of life dimensions: 1) physical well-being (5 items), 2) psychological well-being (7 items), 3) parents/guardians relations & autonomy (7 items), 4) social support & peers (4 items), and 5) school environment (5 items).
  The questions are answered on a 5-point likert scale. Scores can be created for each of the five dimensions. The methodology given in the developers manual will be used to obtain the T-scores; mean (±SD) scores of 50 ± 10 define normality for children and adolescents aged 8-18 years across Europe. Higher scores indicate a better health-related quality of life.
The adolescents domain specific self-evaluation of competence or adequacy | Measured baseline and after 12 months
  Assessed through Harter's Self-perception Profile for Adolescents (SPPA). The instrument consists of seven subscales covering the following domains: 1) scholastic competence, 2) social competence, 3) athletic competence, 4) physical appearance, 5) job competence, 6) close friendship, and 7) romantic appeal.
  Each subscale contains four items, each having four options: 1 (Describes me very poorly), 2 (Describes me fairly poorly), 3 (Describes me fairly well), and 4 (Describes me very well), providing a mean score of perceived competence in that area, ranging from 1 (lowest level of self-esteem) to 4 (highest level of self-esteem).
Symptoms of anxiety and depression | Measured baseline and after 12 months
  Assessed by the short version of Hopkins Symptom Checklist (HSCL-10). HSCL-10 consists of 10 symptoms or problems that people sometimes have in which adolescents answered how much the symptoms have bothered or distressed them during the last week.
  All 10 questions have 4 response categories: 'Not at all', 'A little', 'Quite a bit' and 'Extremely'. The responses are summarized across all items and the mean score is used as a measure of psychological distress. Higher values indicates higher psychological distress.
Learning environment in the classroom | Measured baseline and after 12 months
  The Classroom Climate Scale is used to assess learning environment. This instrument consist of 22 questions related to intrinsic and extrinsic motivation, anticipation and teacher-student relations.
  All questions are answered on a four-point scale: "Strongly agree", "Somewhat agree", "Somewhat disagree", "Strongly disagree". All points are summed to a total score. Higher scores indicates higher classroom environment.
School environment | Measured baseline and after 12 months
  Learning environment at school in general is self-reported in a questionnaire. It consist of three separate questions, and the questions are answered on a 7-point likert scale ranging from "totally disagree" to "totally agree". A mean score from the three questions will be made, and a higher score indicates better school environment.

OTHER OUTCOMES:
Body mass index | Measured baseline and after 12 months
  Body mass (weight; 0.1 kg) is measured using an electronic scale with participants wearing light clothing. Stature (height; 0.1 cm) is measured using a portable stadiometer. The individual face forward, with shoes removed. Body mass index is calculated as body weight (kg) divided by the height squared (m2).
Waist circumference | Measured baseline and after 12 months
  Measured with an ergonomic circumference measuring tape. The measure is taken at the midway between the lower rib and iliac crest with the individual's abdomen relaxed at the end of a gentle expiration.
Satisfaction of basic psychological needs | Measured baseline and after 12 months
  Assessed by Basic Psychological Needs in Exercise Scale (BPNES). BPNES consist of 12 questions that are answered on a 7-point Likert scale (ranging from 1 (Certainly untrue) to 7 (Certainly true)). The responses are summarized and a mean score is made. Higher values indicates higher satisfaction.
Emotional responses to physical education | Measured baseline and after 12 months
  Assessed by the Basic Emotions Trait Test (BETT). BETT consists of 9 statements that will measure positive, negative and eudaimonic emotions. Participants respond on a 7-point Likert scale ranging from 1 (Never) to 7 (Always). The responses are summarized across the three sub-scales and a mean score for each sub-scale is made. Higher values indicates higher emotions.
Eagerness to join physical education | Measured baseline and after 12 months
  Assessed by Eagerness for Physical Activity Scale (EPAS). EPAS is a one-dimensional scale, consisting of 12 statements that affect emotional expressions and cognitive assessments as well as future physical activity behavior. The participants respond to the statements on a scale ranging from 1 (completely disagree) to 7 (completely agree). The responses are summarized and a mean score is made. Higher values indicates higher eagerness.

CONTACTS AND LOCATIONS:
Overall Officials: Elin Kolle, PhD, Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 24 months of study completion
Access Criteria: Data access will be reviewed by the study's publication group. Requestors will be required to sign a data access agreement

REFERENCES:
- [Derived] Malnes L, Haugen T, Nordbo ECA, Ivarsson A, Kolle E, Resaland GK, Solberg RB, Avitsland A, Berntsen S. Objectively measured environmental factors in relation to school travel mode among adolescents: a decision tree analysis. Int J Behav Nutr Phys Act. 2025 Mar 4;22(1):26. doi: 10.1186/s12966-025-01727-6. PMID 40038743
- [Derived] Malnes L, Berntsen S, Kolle E, Ivarsson A, Dyrstad SM, Resaland GK, Solberg R, Haugen T. School-based physical activity in relation to active travel - a cluster randomized controlled trial among adolescents enrolled in the school in motion study in Norway. Int J Behav Nutr Phys Act. 2023 Nov 21;20(1):136. doi: 10.1186/s12966-023-01534-x. PMID 37990252
- [Derived] Leibinger E, Avitsland A, Resaland GK, Solberg RB, Kolle E, Dyrstad SM. Relationship between health-related quality of life and physical fitness in Norwegian adolescents. Qual Life Res. 2023 Apr;32(4):1133-1141. doi: 10.1007/s11136-022-03309-6. Epub 2022 Dec 17. PMID 36527570
- [Derived] Malnes L, Haugen T, Hansen BH, Kolle E, Berntsen S. Establishing the Convergent Validity of the Travel Habit Questions in the Health Behavior in School-Aged Children Questionnaire by Quantifying Active Travel in Norwegian Adolescents. Front Sports Act Living. 2022 Apr 6;4:761723. doi: 10.3389/fspor.2022.761723. eCollection 2022. PMID 35463834
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Solberg RB, Steene-Johannessen J, Anderssen SA, Ekelund U, Safvenbom R, Haugen T, Berntsen S, Avitsland A, Lerum O, Resaland GK, Kolle E. Effects of a school-based physical activity intervention on academic performance in 14-year old adolescents: a cluster randomized controlled trial - the School in Motion study. BMC Public Health. 2021 May 6;21(1):871. doi: 10.1186/s12889-021-10901-x. PMID 33957895
- [Derived] Kolle E, Solberg RB, Safvenbom R, Dyrstad SM, Berntsen S, Resaland GK, Ekelund U, Anderssen SA, Steene-Johannessen J, Grydeland M. The effect of a school-based intervention on physical activity, cardiorespiratory fitness and muscle strength: the School in Motion cluster randomized trial. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):154. doi: 10.1186/s12966-020-01060-0. PMID 33243246
- [Derived] Avitsland A, Leibinger E, Haugen T, Lerum O, Solberg RB, Kolle E, Dyrstad SM. The association between physical fitness and mental health in Norwegian adolescents. BMC Public Health. 2020 May 24;20(1):776. doi: 10.1186/s12889-020-08936-7. PMID 32448149

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03817047/Prot_SAP_001.pdf